CLINICAL TRIAL: NCT06055400
Title: Ultrasound-guided Interventions With Augmented Reality Visualization: A Randomized Crossover Study Investigating Trainees' Performance and Cognitive Load During Skill Acquisition
Brief Title: An Investigation of Trainees' Performance in Augmented Reality Simulation for Invasive Procedure Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shu-Chen Liao (Other)
Responsible Party: Sponsor-Investigator, Shu-Chen Liao, Director of simulation center, Principal Investigator, Clinical Associate Professor., Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CGMH AR
Record Dates: First submitted 2023-09-06; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: Cognitive load; Clinical competence; Augmented reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard US (No Intervention): The participants underwent CVC placement using standard ultrasound guidance.
- AR-US (Experimental): The participants underwent CVC placement using AR-HMD ultrasound guidance.
  Interventions: Device: AR-US

INTERVENTIONS:
Device: AR-US — The ultrasound imagery is projected onto the glasses, and participants use the AR-US throughout the entire CVC placement procedure
  Other Names: augmented reality smart glasses
  Arms: AR-US

SUMMARY:
The primary aim of this study is to measure the efficacy of augmented reality technology in ultrasound-guided medical intervention.

DETAILED DESCRIPTION:
BACKGROUND: A significant challenge facing novice physicians is mastering ultrasound(US)-guided procedures, such as central venous catheter (CVC) placement. CVC placements are typically performed on critically ill patients and demand precision and speed. Physicians are often required to switch focus between the ultrasound screen and the patient, memorize multiple images, coordinate hand-eye movements, and interpret 2D images in a 3D context simultaneously. These complexities pose challenges in spatial orientation and impose a considerable cognitive load, affecting both learning and performance. Within the pedagogical landscape, medical educators are exploring the potential merits of Augmented Reality (AR) via head-mounted displays to enhance immersive learning experiences in clinical settings. This study aimed to determine whether AR could ease challenges related to spatial orientation and cognitive overload during this procedure and ultimately enhance skill acquisition for trainees.

Intervention:

Prior to the commencement of the trial, all participants verified their previous training in ultrasound-guided CVC placement. They also provided their written informed consent. The participants are set to be split into two groups as part of a crossover design: the first group will initially be subjected to the traditional ultrasound-guided CVC placement, whereas the second group will begin with the AR-assisted CVC placement

STUDY IMPLICATIONS:

Leveraging AR technology in skill acquisition may reduce trainees' cognitive burden and improve trainee efficiency during ultrasound-guided CVC placement procedures..

ELIGIBILITY:
Inclusion criteria

1. Age greater than or equal to 20 years
2. Final-year medical students (UGY)
3. Post-year graduate physicians (PGY)
4. Physicians who have previously received training in ultrasound-guided CVC placement or who have experience with such procedures.

Exclusion Criteria:

Participants who experience discomfort during the process, are pregnant, have high blood pressure, have experienced recent dizziness, have inner ear diseases, suffer from claustrophobia, have undergone recent surgery, have visual impairment, have heart disease, have epilepsy, or refuse to participate.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Performance of CVC Placement | up to 30 minutes
  first pass rate in percent, success/failure rate in percent, number of attempts, number of artery punctures, the number of operator head turns in counts, venous access time (from start to venous access in seconds), lag time (from access ultrasound probe to venous access in seconds), catheterization time (from start to complete catheterization in seconds), total time in seconds.

SECONDARY OUTCOMES:
Cognitive load of CVC placement | up to 30 minutes
  Cognitive load of CVC placement measured in NASA Task Load Index. The score of the NASA task load index ranges from 0 to 20. A higher score indicates a higher cognitive load.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Chen Liao, M.D., Principal Investigator — Department of Emergency Medicine, Keelung Chang Gung Memorial Hospital, Keelung, Taiwan.
Locations (1):
- Keelung Chang Gung Memorial Hospita, Keelung, Guishan Dist., Taiwan

REFERENCES:
- [Derived] Liao SC, Shao SC, Gao SY, Lai EC. Augmented reality visualization for ultrasound-guided interventions: a pilot randomized crossover trial to assess trainee performance and cognitive load. BMC Med Educ. 2024 Sep 27;24(1):1058. doi: 10.1186/s12909-024-05998-8. PMID 39334275